CLINICAL TRIAL: NCT04745182
Title: A Tailored Program to Promote Well-being and Physical Activity in Mid-life Adults With Low Physical Activity
Acronym: MASTERY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jeff C. Huffman, MD, Director, Cardiac Psychiatry Research Program, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2019P002328
Record Dates: First submitted 2021-02-02; First posted 2021-02-09 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Middle Aged; Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: All participants were in the same group and received the same intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MASTERY (Experimental): For each session, a PP exercise will be described in the manual, with instructions and space to write about the exercise and its effects. Next, an MI section will outline specific MI-based topics (e.g., pros/cons, managing slips) and will contain space to write a specific physical activity goal and to track physical activity (e.g., through step counter data) over the subsequent week. At the in-person visit #2, interventionists will explain PP exercise 1 and MI session 1 to the participants. Calls will last ~30 minutes. Participants will then independently complete PP exercises and MI-based goals and review them at phone sessions over 12 weeks. PP and MI components will be delivered stepwise within sessions (rather than intertwined) based on our experience, participant feedback, and pilot work.
  Interventions: Behavioral: MASTERY

INTERVENTIONS:
Behavioral: MASTERY — A 12-week, phone-delivered intervention utilizing positive psychology (PP), motivational interviewing (MI), and specific midlife modules (e.g., on time management, financial stress, caregiving stress, or occupational stress) to promote physical activity and well-being in mid-life adults.

SUMMARY:
This is a single-arm pilot trial to examine the feasibility, acceptability, and preliminary efficacy of the 12-week, phone-delivered, Midlife Activity, Stress reduction, Time Efficiency, Resilience, and Youthfulness (MASTERY) intervention, which utilizes positive psychology (PP), motivational interviewing (MI), and specific midlife modules (e.g., on time management, financial stress, caregiving stress, or occupational stress) to promote well-being and physical activity in mid-life adults.

DETAILED DESCRIPTION:
This is a single-arm proof-of-concept trial of a phone-delivered positive psychology-motivational interviewing (PP-MI) intervention, with content adapted to midlife persons. Midlife adults with low physical activity were recruited from outpatient clinics, completed baseline outcome measures (including wearing an accelerometer to measure activity for one week), completed the 12-week MASTERY intervention, and then completed a follow-up session to obtain repeat outcome information. The intervention, which involved weekly phone sessions with a trained study team member, included the completion of PP exercises, setting physical activity goals, and completion of activities to reduce midlife-specific stressors. The primary outcomes were feasibility and acceptability, and secondary outcomes included accelerometer-measured physical activity and self-report outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age 45-64 years at time of enrollment.
* Low physical activity (defined as ≤150 minutes/week of MVPA, in accordance with consensus recommendations for moderate or greater intensity aerobic physical activity and measured using a brief version of the well-validated International Physical Activity Questionnaire (IPAQ) scale.

Exclusion Criteria:

* Existing coronary artery disease. Coronary artery disease will be identified through review of the medical record, with clarification by participants' primary clinician if needed, as part of recruitment procedures. Existing coronary artery disease will be defined as a prior acute coronary syndrome (unstable angina or myocardial infarction) or diagnosed via cardiac catheterization.
* To meet criteria for a prior acute coronary syndrome, for myocardial infarction, patients must have experienced at least two of three World Health Organization criteria for an acute myocardial infarction: typical chest pain, elevated cardiac enzymes, and electrocardiographic changes consistent with myocardial infarction.
* For unstable angina, participants must have had new onset angina within 2 months, exacerbation of previous angina with rest pain or with minimal exercise, or angina within 2 weeks of myocardial infarction, with confirmation of this diagnosis by the patient's primary medical provider or inpatient treatment team; this definition has been used in prior trials.
* To meet criteria for coronary artery disease diagnosed at cardiac catheterization, participants must have had 50% stenosis of the left main artery or 70% stenosis of another coronary artery, consistent with consensus definitions of obstructive coronary artery disease.
* Cognitive disturbance precluding participation or informed consent, as identified using a six-item cognitive screen designed to assess suitability for research participation.
* Lack of available telephone.
* An inability to communicate in English.
* A condition limiting physical activity (e.g., arthritis, chronic obstructive pulmonary disease), identified by patient and medical record, confirmed by primary medical provider as needed.
* Participation in similar programs (e.g., mind-body interventions) as reported by patients.

Ages: 45 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-03-19 (Actual); Study Completion 2020-03-19 (Actual)

PRIMARY OUTCOMES:
Proportion of total phone sessions completed | 12 weeks
  To assess the feasibility of the intervention
Mean ease ratings of exercises | 12 weeks
  To assess how easy participants found the assigned exercises. Ratings will be made on a scale of 0-10, with 0 being very difficult and 10 being very easy.
Mean utility ratings of exercises | 12 weeks
  To assess how useful participants found the assigned exercises. Ratings will be made on a scale of 0-10, with 0 being not at all useful and 10 being very useful.

SECONDARY OUTCOMES:
Proportion of sessions completed by participants | 12 weeks
  To assess the feasibility of study procedures. We will divide the number of phone sessions completed by participants by the total number of phone sessions that could have been completed.
Change in Moderate-Vigorous Physical Activity | Change from Baseline to 12 weeks
  ActiGraph GT3X+ step counters are validated as measures of physical activity and have been used in numerous studies of physical activity in patients with medical illness. In this trial, participants will wear the accelerometer for one week at baseline and at 12 weeks. We will report change from baseline to 12 weeks in the average number of minutes of MVPA performed per day.
Change in Positive Affect | Change in score from Baseline to 12 weeks
  The positive affect items on the Positive and Negative Affect Schedule (PANAS), a well-validated scale used in other intervention trials and in patients with medical illnesses, will be used to measure positive affect (Range: 10-50). Change will be calculated by subtracting the score at baseline from the score at 12 weeks. Higher scores indicate higher levels of positive affect.
Change in Optimism | Change in score from Baseline to 12 weeks
  Life Orientation Test-Revised is a well-validated 6-item instrument used to measure dispositional optimism (Range: 0-24). Change will be calculated by subtracting the score at baseline from the score at 12 weeks. Higher scores indicate higher levels of optimism.
Change in Depression | Change in score from Baseline to 12 weeks
  The Hospital Anxiety and Depression Scale (HADS)-depression subscale will be used to measure depression. This is a well-validated scale with few somatic symptom items that can confound mood/anxiety assessment in medically-ill patients (Range: 0-21). Change will be calculated by subtracting the score at baseline from the score at 12 weeks. Higher scores indicate higher levels of depression.
Change in Anxiety | Change in score from Baseline to 12 weeks
  The Hospital Anxiety and Depression Scale (HADS)-anxiety subscale will be used to measure anxiety. This is a well-validated scale with few somatic symptom items that can confound mood/anxiety assessment in medically-ill patients (Range: 0-21). Change will be calculated by subtracting the score at baseline from the score at 12 weeks. Higher scores indicate higher levels of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Jeff C Huffman, MD, Study Director — Massachusetts General Hopsital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huffman JC, Massey CN, Chung WJ, Harnedy LE, Carrillo A, Feig EH, Celano CM. A Psychological-Behavioral Intervention to Improve Physical Activity in Midlife Adults With Low Baseline Physical Activity. Prim Care Companion CNS Disord. 2021 Jul 29;23(4):20m02876. doi: 10.4088/PCC.20m02876. PMID 34324798